CLINICAL TRIAL: NCT03820973
Title: Development and Pilot Testing of Video-based Deliver of Brief Cognitive Behavioral Therapy for Anxiety
Brief Title: Brief Cognitive Behavioral Therapy for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Cully, Clinicial Research Psychologist, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-44258
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Anxiety
Keywords: brief Cognitive Behavioral Therapy; VA Video Connect to home
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief CBT for Anxiety (Experimental): Participants will receive Brief Cognitive Behavioral Therapy for Anxiety (bCBT). Sessions with clinicians will be provided via VA Video Connect to Home (VVC-H). Participants will have the option to select from a list of skills to tailor to his/her preferences. Participants will be able to receive up to 9 total sessions and generally last 30 to 40 minutes. For the purpose of this study, treatment duration will be limited to 3 months to ensure standardization of study outcome measures.
  Interventions: Behavioral: Brief CBT for Anxiety

INTERVENTIONS:
Behavioral: Brief CBT for Anxiety — All participants will receive psychoeducation on anxiety and bCBT treatment approach, work on setting goals, begin self-monitoring, and select skill sessions that fit his/her most pressing needs. Available skills: Relaxation-Diaphragmatic breathing is a simple relaxation technique that increases oxygen flow and reduces the unpleasant physiological sensations associated with anxiety; Exposure - designed to educate Veterans about the role of avoidance in maintaining anxiety problems, as well as information about how to reduce avoidance through exposure exercises; Cognitive - Veterans may opt to address anxiety and worry through modifying negative thinking patterns. Two available options - Increasing Helpful Thoughts and Managing Unhelpful Thoughts.

SUMMARY:
The proposed clinical intervention is a modular skills-based intervention for flexible delivery of care, measurement-based care practices, and integration of exposure strategies critical for anxiety symptom reduction. Notably, the treatment targets anxiety symptoms rather than diagnoses to improve use in PCMHI and CBOC settings. The pilot study will develop and conduct preliminary testing of bCBT for anxiety using Veterans Affairs (VA) Video Connect to Home (VVC-H) to deliver care.

DETAILED DESCRIPTION:
Anxiety disorders are identified in over 30% of primary care patients and are associated with substantial functional impairment, poor health-related quality of life, and suicide; however, rates of treatment are low. In contrast to advances in improving treatment of depression and posttraumatic stress disorder in VA, far less attention has been given to anxiety disorders. In the absence of VA clinical practice guidelines for anxiety disorders, evidence-based treatment practices are unstandardized in VA primary care and Community Based Outpatient Clinics (CBOCs). Cognitive behavioral therapy (CBT) is an evidence-based intervention for the anxiety disorders but was developed for use in specialty mental health settings and often targets individual anxiety disorders (e.g.generalized anxiety, panic, and social phobia) with diagnosis-specific treatment packages. These interventions are not practical for primary care and CBOC settings where treatment must be brief and focused on reduction of anxiety symptoms rather than targeted anxiety diagnoses. Further complicating the delivery of CBT for anxiety disorders is that repeated exposure to feared cues is considered a critical component of CBT for anxiety but is rarely used in these settings. Providers within VA currently have no standardized options for delivering brief evidence-based psychotherapy for Veterans with anxiety. Although Primary Care Mental Health Integration (PCMHI) and CBOCs increase access to mental health services, VA recognizes the need to deliver mental health services using video to home technology to increase access, decrease barriers (i.e., geographic distance, transportation, travel time, stigma, child care) and provide more Veteran-centric care. VA is pioneering implementation of VA Video Connect to Home (VVC-H) technology in specialty mental health clinics, but VVC-H continues to be rarely used and little is known about the implementation potential of VVC-H to improve psychotherapy access and outcomes in primary care and CBOC settings. In summary, VA needs a flexible evidence-based approach for anxiety that fits within primary care and CBOC settings and offers innovative delivery strategies to increase access to care. Although treatment in PCMHI and CBOC settings must be time-limited, it must also be highly effective. The investigators have developed robust brief CBT (bCBT) interventions and provider support programs for depression and is now seeking to address anxiety using a similar approach. The proposed clinical intervention will use state-of-the-art practices including delivery of services via VVC-H. This open trial seeks to recruit 12 Veterans who have significant anxiety symptoms according to the GAD-7 (standard assessment tool for VA clinical settings). Veterans will be recruited from the Michael E. DeBakey VAMC primary care clinic and affiliated Community Based Outpatient Clinics (CBOCs).

ELIGIBILITY:
Inclusion Criteria:

Veteran participants: The sample will include Veterans who:

1. receive care at the Houston VA and surrounding area CBOCs,
2. have documentation in the medical chart of an anxiety disorder or anxiety-related problems, and
3. report clinically significant symptoms of anxiety, defined as a score of 10 or greater on the Generalized Anxiety Disorder Scale, 7th edition (GAD-7).

Exclusion Criteria:

Veteran participants will be excluded for factors that would render bCBT inappropriate, including:

1. cognitive impairment;
2. presence of bipolar, psychotic or substance use disorders, and
3. Veteran is currently receiving psychotherapy for anxiety. If receiving medications that target anxiety Veterans WILL NOT be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder - 7 item scale - looking at change in scores over time | Baseline, and 3-Months
  scale used to measure anxiety, scores range from 0 to 21, where higher scores equal higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cully, PhD, Principal Investigator — Michael E. DeBakey VAMC
Locations (1):
- Michael E. DeBakey VAMC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No